CLINICAL TRIAL: NCT06997783
Title: Acute Effects of Moderate and Maximal Squat Loading
Brief Title: Acute Effects of Moderate and Maximal Squat Loading on Ju-do-Specific Performance in Elite Judokas
Status: Completed | Type: Observational
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: İnönü University (Unknown)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Other Study IDs: PNU2
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard Warm-Up (SWU):: This condition will involve a typical judo-specific warm-up protocol lasting approximately 25 minutes. It will include:
  8-10 minutes of mobility and dynamic flexibility exercises focusing on major joints and muscle groups (e.g., hip circles, arm swings, and leg kicks)
  Interventions: Other: warm up
- A moderate-load PAPE warm-up (80% of 6-repetition maximum): This experimental warm-up condition will consist of the same initial exercises as the SWU, followed by the addition of a moderate-load squat-based PAPE protocol. The structure will include: Back squats performed at 80% of the participant's 6-repetition maximum (6RM)
  3 sets of 3 repetitions, performed with maximal effort and proper form, under supervision
  Rest intervals of 3-5 minutes between sets to allow partial recovery and facilitate potentiation.
  Interventions: Other: warm up
- A maximal-load PAPE warm-up (100% of 1-repetition maximum): This condition will also begin with the same general and judo-specific exercises as the SWU, followed by a high-intensity PAPE protocol:
  Extended rest periods of 4-5 minutes between the final lift and performance testing to minimize fatigue effects The full warm-up will also be completed within a 25-minute session
  Interventions: Other: warm up

INTERVENTIONS:
Other: warm up — 1. Standard Warm-Up (SWU):
     This condition will involve a typical judo-specific warm-up protocol lasting approximately 25 minutes.
  2. Moderate-Load PAPE Warm-Up (80% of 6RM):
     This experimental warm-up condition will consist of the same initial exercises as the SWU, followed by the addition of a moderate-load squat-based PAPE protocol.
  3. Maximal-Load PAPE Warm-Up (100% of 1RM):
  This condition will also begin with the same general and judo-specific exercises as the SWU, followed by a high-intensity PAPE protocol: 1-2 sets of a single repetition of back squats at 100% of the participant's 1-repetition maximum (1RM).

SUMMARY:
This study will investigate the acute effects of two squat-based post-activation performance enhancement (PAPE) protocols-moderate load (80% of 6RM) and maximal load (100% of 1RM)-on judo-specific performance in elite male judokas. A total of 20 national-level male judokas will participate in a randomized, counterbalanced protocol across a 3-week period. Each participant will complete standard and experimental warm-up sessions followed by the Special Judo Fitness Test. Outcome measures will include total throws, immediate and 1-minute post-exercise heart rates, and the performance index. The study aims to determine the optimal PAPE intensity for enhancing performance while minimizing fatigue in combat sport athletes.

DETAILED DESCRIPTION:
This study will examine the acute effects of two different squat-based post-activation performance enhancement (PAPE) protocols on judo-specific performance in elite male judokas. The purpose is to identify an optimal loading strategy that enhances performance without inducing excessive fatigue, which is critical for pre-competition preparation in combat sports.

A total of 20 male judokas with at least two years of competitive experience at the national level will be recruited. Participants will undergo three different warm-up conditions in a randomized, counterbalanced order over a 3-week period:

A standard warm-up (SWU) based on typical judo routines

A moderate-load PAPE warm-up (80% of 6-repetition maximum)

A maximal-load PAPE warm-up (100% of 1-repetition maximum)

Each warm-up session will last approximately 25 minutes. After each warm-up, participants will perform the Special Judo Fitness Test (SJFT), which assesses anaerobic capacity, throwing ability, and recovery. Outcome measures will include the number of total throws, immediate and 1-minute post-test heart rate, and the SJFT performance index.

It is expected that the moderate-load (80%) PAPE protocol will yield the greatest improvements in judo-specific performance, offering a better balance between muscle potentiation and fatigue than the maximal-load (100%) or standard warm-up conditions. These findings will inform practical warm-up strategies for combat sport athletes aiming to enhance performance immediately before competition.

ELIGIBILITY:
Inclusion Criteria:

* Male judokas aged 18-25 years
* Minimum of 2 years of continuous judo training experience
* Active participation in national-level judo competitions
* Free from injury for at least 6 months prior to the study
* Able to perform high-intensity resistance and sport-specific exercises
* Willing to participate and provide informed consent

Exclusion Criteria:

* Current musculoskeletal injury or medical condition affecting performance
* History of surgery within the last 6 months
* Cardiovascular, respiratory, or neurological conditions contraindicating intense physical activity
* Use of medications that affect muscle performance or recovery
* Participation in other performance-enhancement or warm-up research studies during the study period
* Inability to follow study instructions or complete testing protocols

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of elite male judokas aged 18 to 25 years who have a minimum of two years of continuous judo training experience and are actively competing at the national level. Participants will be recruited from local judo clubs and training centers. All individuals must be in good health, free from recent injuries, and capable of performing high-intensity strength and sport-specific exercises. The sample will represent a homogenous group of trained athletes, enabling a focused investigation of post-activation performance enhancement (PAPE) protocols on judo-specific performance outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Special Judo Fitness Test (SJFT). | Immediately post-intervention on Day 1, Day 8, and Day 15 (across the 3-week study period)
  The SJFT will be used to assess judo-specific performance through repeated throwing efforts within defined time intervals. The test consists of three periods of activity (15 seconds, 30 seconds, and 30 seconds) separated by 10-second rest intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided